CLINICAL TRIAL: NCT04083547
Title: Cirkulerande Tumörceller Hos Patienter Med Bukhinnespridda tumörer
Brief Title: Circulating Tumour Cells in Patients With Peritoneal Metastases
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC study
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Circulating Tumor Cell; Peritoneal Metastases; Hyperthermic Intraperitoneal Chemotherapy
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIPEC group: All patients undergoing HIPEC will asked to join this prospective study.
  Interventions: Diagnostic Test: iCellate

INTERVENTIONS:
Diagnostic Test: iCellate — New method of circulating tumour cell detection and capture.

SUMMARY:
This study aims to evaluate the prognostic value of circulating tumour cells (CTC) in patients undergoing cytoreductive surgery and hyperthermic intraperitoneal chemotherapy due to gastrointestinal cancers that have spread to the peritoneum.

DETAILED DESCRIPTION:
CTCs har extracted by way of a new method at baseline, during surgery, and postoperatively. The occurence of such CTCs will be investigated for prognostic evaluation. Patients will be follow-up by Clinical routine. Disease recurrence and overall survival will be the endpoint used.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal metastases being treated with cytoreductive surgery and hyperthermic intraperitoneal chemotherapy

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients being treated in Uppsala with CRS and HIPEC will be asked to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Prognostic value | 2 year.
  Prediction of survival and recurrence according to the occurrence of CTCs.

CONTACTS AND LOCATIONS:
Locations (1):
- Akademiska Sjukhuset (Uppsala University hospital), Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided